CLINICAL TRIAL: NCT03127345
Title: Omega 3 Fatty Acid Treatment for Pediatric Musculoskeletal Health
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Melissa Putman, Attending in Endocrinology, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-P00024279
Record Dates: First submitted 2017-04-07; First posted 2017-04-25 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Esophageal Atresia
MeSH Terms: conditions — Esophageal Atresia | interventions — fish oil triglycerides; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omegaven (Experimental): 15 infants with esophageal atresia undergoing surgical repair will receive Omegaven 1 g/kg/day IV infused over 8-24 hours for 28 days
  Interventions: Drug: Omegaven
- Intralipid (Active Comparator): 15 infants with esophageal atresia undergoing surgical repair will receive the standard of care lipid formulation (Intralipid) as per hospital protocol for 28 days
  Interventions: Drug: Intralipid

INTERVENTIONS:
Drug: Omegaven — Intravenous omega 3 fatty acid administration
  Arms: Omegaven
Drug: Intralipid — Standard of care
  Arms: Intralipid

SUMMARY:
This is a randomized clinical trial comparing Omegaven® treatment with standard of care (soybean-based lipid formulation, Intralipid®) on bone health outcomes in infants with esophageal atresia (EA) undergoing surgical repair at Boston Children's Hospital.

DETAILED DESCRIPTION:
Medical treatments and disease pathophysiology can result in prolonged immobilization that places hospitalized infants and children at risk for serious musculoskeletal complications including bone loss, fragility fractures, and muscle atrophy. Patients at the highest risk for inpatient fracture include premature infants, children with cerebral palsy, spinal cord injury, neuromuscular disorders (e.g., Duchenne Muscular Dystrophy or Spinal Muscular Atrophy), lengthy post-operative immobilization such as esophageal atresia (EA), and prolonged use of parenteral nutrition (PN). These fractures can result in significant discomfort, increase medical costs, may require surgical intervention, and may result in long term deleterious effects on musculoskeletal health.

Omega-3 polyunsaturated fatty acids (O3PuFA) are important bio-mediators modulating bone formation and remodeling. We demonstrated that O3PuFA provide protection of bone microstructure by increasing the number of trabecular elements and subsequently strengthening the trabecular network in young mice. Human studies suggest an association between O3PuFA intake and increased bone mineral density (BMD) in adults, and we also demonstrated decreased fracture risk in infants. O3PuFA may reduce bone resorption by modulating inflammatory cytokines and inhibiting osteoclast differentiation and activity, and may also increase bone formation by increasing osteoblast differentiation and activity, which may provide the explanation for the observed skeletal benefits.

In this study, we propose the use of intravenous O3PuFA (Omegaven® , Fresenius Kabi, Bad Hamburg Germany) administration for the prevention of musculoskeletal complications due to immobilization in infants. Boston Children's Hospital (BCH) has more than 15 years' experience with this O3PuFA product, having treated more than 250 infants and children. Omegaven is currently under review by the FDA for treatment of infants with PN-associated liver disease.

The proposed study is a randomized, double blind clinical trial using comparing Omegaven® administration to the current standard of care (soybean-based lipid formulation, Intralipid®) on musculoskeletal health in high risk infants with EA admitted at BCH. Infants with EA have been observed to have dramatic bone loss and a very high fracture rate (over 40%) related to their prolonged post-operative immobilization; therefore, these patients represent the ideal model to evaluate this intervention. By targeting this particular patient population at such high risk for musculoskeletal complications and limited confounding factors, the effects of our intervention will have the highest probability of being identified if such a benefit does exist.

In this pilot study, thirty-two infants with EA will be randomized to either treatment arm for a four-week treatment period. Safety outcomes will include regular laboratory monitoring as per routine standard of care. Efficacy outcomes will include (1) computed tomography (CT) of the bilateral distal femurs at baseline and at 4 weeks, which will provide skeletal outcomes including volumetric bone density, bone geometry, and bone strength estimates, (2) serum and urine markers of bone turnover, and (3) incidence of fracture in the post-operative period. All subjects will continue to receive treatments according to standard of care regardless of group assignment, including physical therapy, nutritionist consult, fracture precautions, and regular laboratory monitoring per discretion of the primary medical team.

ELIGIBILITY:
Inclusion Criteria:

1) Diagnosis of long-gap EA (esophageal gap length >3cm) 2) Age <12 months (not yet reached 12 month birthday) 3) Anticipated surgical repair for management of EA utilizing esophageal traction requiring prolonged intubation, muscle relaxation, and parenteral nutrition dependence.

1. Known genetic bone disease, including osteogenesis imperfecta, idiopathic infantile hypercalcemia, and vitamin D resistant rickets
2. Prior fragility fracture (including humerus or femur)
3. Anticipated hospital stay of less than 4 weeks (28 days)
4. Impaired lipid metabolism
5. Severe hemorrhagic disorder. This is defined as platelets <50 K cells/uL, hemoglobin <7 g/dL, and INR >2.0. Patients treated with full therapeutic anticoagulation (i.e. for treatment of thrombosis) will also be excluded. This does not include patients on anticoagulants at prophylactic doses.
6. Unstable diabetes mellitus
7. Collapse and shock
8. Stroke/embolism
9. Recent cardiac infarction
10. Undefined coma status
11. Allergy to egg or fish
12. Prior treatment with Omegaven
13. Liver disease (defined as elevated serum aminotransferases and/or direct bilirubin at the time of enrollment)
14. Renal disease (defined as serum creatinine level above the normal range for age at the time of enrollment)
15. Acid or base disorders (defined as serum bicarbonate less than 10 or greater than 40)
16. Preterm infants less than 32 weeks gestation or birthweight <1500 grams who have not had a cranial ultrasound that showed no evidence of intraventricular hemorrhage at 36-40 weeks corrected gestational age
17. Prior diagnosis of intraventricular hemorrhage

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in total volumetric bone mineral density of the distal femur | Baseline and 28 days
  Computed tomography

SECONDARY OUTCOMES:
Cortical and trabecular volumetric bone mineral density of the distal femur | Baseline and 28 days
  Computed tomography
Bone geometry and bone strength estimates of the distal femur | Baseline and 28 days
  Computed tomography
Bone turnover markers | Baseline, 14 days, and 28 days
  Blood and urine testing
Incidence of fracture | 28 days
  Incidence of fracture
Incidence of adverse events | Daily for 28 days
  Incidence of adverse events

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fallon EM, Nazarian A, Nehra D, Pan AH, O'Loughlin AA, Nose V, Puder M. The effect of docosahexaenoic acid on bone microstructure in young mice and bone fracture in neonates. J Surg Res. 2014 Sep;191(1):148-55. doi: 10.1016/j.jss.2014.04.005. Epub 2014 Apr 12. PMID 24793452
- [Background] Le HD, de Meijer VE, Robinson EM, Zurakowski D, Potemkin AK, Arsenault DA, Fallon EM, Malkan A, Bistrian BR, Gura KM, Puder M. Parenteral fish-oil-based lipid emulsion improves fatty acid profiles and lipids in parenteral nutrition-dependent children. Am J Clin Nutr. 2011 Sep;94(3):749-58. doi: 10.3945/ajcn.110.008557. Epub 2011 Jul 20. PMID 21775562
- [Background] Nehra D, Fallon EM, Potemkin AK, Voss SD, Mitchell PD, Valim C, Belfort MB, Bellinger DC, Duggan C, Gura KM, Puder M. A comparison of 2 intravenous lipid emulsions: interim analysis of a randomized controlled trial. JPEN J Parenter Enteral Nutr. 2014 Aug;38(6):693-701. doi: 10.1177/0148607113492549. Epub 2013 Jun 14. PMID 23770843